CLINICAL TRIAL: NCT01169285
Title: Prospective Observational
Brief Title: Efficiency and Efficacy of the Distress Thermometer in the Burn and Wound Population (Research Mentoring High Student Project)
Status: Completed | Type: Observational
Sponsor: Saint Elizabeth Regional Medical Center (Other)
Responsible Party: Pam Wiebelhaus, Saint Elizabeth Regional Burn Center
Other Study IDs: 609-044
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2009-05

CONDITIONS: Burns
Keywords: Burn Department Nursing Staff
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
The purpose of the study is to test the efficiency and efficacy of the Distress Thermometer of patients admitted to the tertiary Burn and Wound Center. The American Cancer Society and the National Comprehensive Cancer Network published treatment guidelines in 2005 adopting the use of the Distress Thermometer as the preferred adjunct assessment tool of a patient's emotional well-being. A literature search provided extension of the tool to a Cardiac Follow-up Clinic. The Distress Thermometer is currently used with oncology patients at Saint Elizabeth.

The emotional well being of patients and their significant others is a hallmark of wholistic care. The simple Likert scale of 0-10 has a trigger for further assessment and/ or intervention at four. The validity testing of the tool was done against the Hospital Anxiety and Depression Scale (HADS) and the Brief Symptom Inventory (BSI-18).

The purpose of this study is to measure the efficiency and efficacy of the documentation of the Distress Thermometer to patients admitted to a tertiary Burn and Wound Care Center. The frequency of the documentation will be counted and type of documentation will be categorized.

ELIGIBILITY:
Inclusion Criteria:

* nursing staff will be nurses working the evening/night shift beginning at 1900.

Exclusion Criteria:

* all patients on the ventilator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Burn Department Nurses and Burn Patients
Sampling Method: Non-Probability Sample
Dates: Start 2009-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)